CLINICAL TRIAL: NCT04682574
Title: Effects of Mega Dose Vitamin C in Critically Ill COVID-19 Patients: A Randomized Control Trial
Brief Title: Role of Mega Dose of Vitamin C in Critical COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Mansoor Hafeez, Doctor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRBEC/BIH/09-2020
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin C (Active Comparator): The dose would be 30 grams a day (10 grams TDS) for 3 days with standard treatment
  Interventions: Drug: Vitamin C
- Placebo (No Intervention): Distill water in the same dose with same standard treatment

INTERVENTIONS:
Drug: Vitamin C — mega dose is given to the selected critically ill patients
  Arms: vitamin C

SUMMARY:
Vitamin C (ascorbic acid) is a water-soluble vitamin having anti-inflammatory, immunomodulatory, anti-oxidative, antithrombotic and antiviral properties. Considering these effects vitamin C should have beneficial impact in patients suffering from sepsis and acute respiratory distress syndrome (ARDS). The current study is designed to assess the beneficial effects of Vitamin C in COVID-19 infected patients.

ELIGIBILITY:
Inclusion Criteria:

critically ill patients admitted in ICU

Exclusion Criteria:

allergic to Vitamin C didnt given the consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Partial pressure of Oxygen in arterial blood to fraction of inspired Oxygen (P/F ratio) | 1 and 4th day
Survival analysis | 28 days follow up

SECONDARY OUTCOMES:
Length of Hospital stay | Admission to discharge
Need for intubation | 28 days
  number of intubations needed in both groups.
Inflammatory markers | before the start of treatment (day 1) and on day 4
  comparison of the inflammatory markers, CRP, D.Dimer, Procalcitonin, LDH, TLC and hematological variables at day four after the intervention started.
APACHE II score | before the start of treatment (day 1) and on day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria Town International Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided